CLINICAL TRIAL: NCT00797537
Title: Concordance Entre l'échographie du Genou et la Radiographie Standard Dans la détection Des Calcifications Dans le Cadre de la Chondrocalcinose Articulaire
Brief Title: Ultrasound and X-ray in Detecting Articular Cartilage Calcification
Acronym: chondro
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: CHU de Limoges, CHU de Limoges
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: I07027/chondrocalcinose
Record Dates: First submitted 2008-11-20; First posted 2008-11-25 (Estimated); Last update posted 2010-09-06 (Estimated); Status verified 2010-09

CONDITIONS: Chondrocalcinosis; Articular Cartilage Calcification
Keywords: Inflammation of bone and cartilage
MeSH Terms: conditions — Chondrocalcinosis; Osteitis | interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Echography — Echography

SUMMARY:
Prospective study with an echography of the 2 knees and radiography of the 2 knees (front and profile) for each patient. If found calcification on ultrasound further examination with ultrasound wrists, hips and shoulders.

DETAILED DESCRIPTION:
Osteo-articular echography is currently recognized as an important development among rheumatologists.

Chondrocalcinosis, which can promote joint inflammation and cartilage degeneration, is highly prevalent in elderly subjects.

Osteo-articular echography is currently reconized as an important development among rheumatologists and can efficiently use to detect Chondrocalcinosis.

The aim of this study is to find a correlation between radiography and echography in detecting CPPD crystal deposition, on a sample of patients and more important with a new generation of ultrasound with a probe superficial performance.

166 patients will be enrolled in this trial and an echography and a radiography of the 2 knees (front and profile) will be done for each patient.

Ih the echography show a calcification, further exams with wrists, hips shoulders echographies will be conducted.

In case of liquid epanchement, analysis of the liquid will be carried in order to eliminate the differential diagnostic including septic arthritis

ELIGIBILITY:
Inclusion Criteria:

* patient> 70 years
* articular pathology of the knee
* consent signed

Exclusion Criteria:

* Not covered by social security

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2008-05; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Knee calcification detected by echography and radiography | Day 1

SECONDARY OUTCOMES:
Calcification description and other localisations finding | Day 1

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Rhumatologie, Limoges, France